CLINICAL TRIAL: NCT05767580
Title: Comparison of Dual Assignment, Cadence, and Gait Speed in Alzheimer's Dementia and Healthy Geriatric Individuals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Senanur AK, Physiotherapist, Kırıkkale University
Other Study IDs: KırıkkaleUniversity-FTR-SA-71
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Dementia
Keywords: dual task; cadance; gait speed; alzheimer demantia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alzehimer demantia geriatric: It is a group of individuals over the age of 65, diagnosed with Alzheimer's dementia, able to walk independently, have no communication problems, and volunteer to participate in the research.
  Interventions: Other: evaluation
- healty geriatric: This is a group of healthy geriatric individuals over the age of 65 who have not been diagnosed with Alzheimer's dementia, can walk independently, have no communication problems, and volunteered to participate in the study.
  Interventions: Other: evaluation

INTERVENTIONS:
Other: evaluation — The Timed Get Up and Go test to assess dual-tasking, the 4m Walk Test to assess gait, and the Footprint Method to assess cadence

SUMMARY:
Tests will be performed in individuals with Alzheimer's dementia to compare dual-task and gait with healthy geriatric individuals.

DETAILED DESCRIPTION:
In this study, it was aimed to compare double assignment, cadence and walking speed in Alzheimer's Dementia and Healthy Geriatric Individuals.

Individuals who can walk independently and who are diagnosed with Alzheimer's Dementia over the age of 65 and healthy individuals will be included in the study. It will be done with 50 people who voluntarily participated in the research.

As a data collection tool; The demographics formula with patient descriptive features is the Timed Get Up and Walk test to turn off double assignment, the 2 Minute Walk Test to evaluate the advertisement, and the Footprint Method to use cadence. It will be assessed with the Mini Mental State Test and the Montreal Cognitive Assessment Test to examine discriminative units.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older,
* Who volunteered to participate in the research,
* Able to walk independently,
* He was diagnosed with Alzheimer's by a physician for the experimental group,
* Having not been diagnosed with Alzheimer's for the control group
* Individuals who have not undergone surgery in the last 6 months
* Individuals who do not have cooperation and communication problems.

Exclusion Criteria:

* Under age 65
* Individuals who do not agree to participate in the research,
* Individuals who have a disability to do physical activity,
* Individuals who have undergone an operation in the last 6 months,
* Individuals with problems of cooperation and communication

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: a total of 50 individuals, including 25 geraitric individuals with Alzheimer's dementia over the age of 65 and 25 healthy geraitric individuals
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-21 (Estimated)

PRIMARY OUTCOMES:
Time Up Go | 6 month
  Timed Start and Continue Test, In the TUG test, individuals stand up from the chair, walk 3 m, walk and sit on a swivel chair. The starting position is standardized with patients feet flat on the floor and their arms resting on the chair. The person is instructed to complete the test at their own pace and as quickly as possible. The test is started with the 'start' command. It ends with him sitting back in the chair. The test is done three times. A 2-minute rest break is given between each trial. The clinician records performance with a stopwatch for each trial.

SECONDARY OUTCOMES:
Dual tasking | 6 month
  Dual tasking (DT) is an experimental neuro-physiological process that requires an individual to perform two tasks simultaneously. When the two activities are done together, the deterioration in the performance of the tasks is defined as Dual Task Deficiency. The formula "DTD = [DT - ST]/TG × 100" was used to calculate the changes in task performances and to determine the deficiency rate, and the results were interpreted proportionally.
Footprint method | 6 month
  The footprint method is carried out by pouring powder in an area of 10 m. Evaluations are made in the middle area of 6 m. The subjects started walking with the left foot and the distances of the sixth, seventh and eighth steps were measured in meters.
Two-Minute Walk Test | 6 month
  Two-Minute Walk Test: It is a test used to evaluate the treatment response in moderately severe heart or lung disease or to evaluate the functional capacity of the person, which is a determinant of mortality and morbidity with a one-time measurement. Reliability, validity and responsiveness of the 2-minute walk test Amy SY Leung , Kam Keung Chan , Kevin Sykes, KS Chan demonstrated in 2006 that the 2MWT is a reliable and valid test for the assessment of exercise capacity and post-rehabilitation response in patients with moderate-to-severe COPD.